CLINICAL TRIAL: NCT03837002
Title: Effect of The Foot Care Protocol Applied to Elderly People on Foot Health Problems and Foot Care Behaviors
Brief Title: Effect of The Foot Care Protocol Applied to Elderly People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Collaborators: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Aslıhan ÇATIKER, Principal Investigator, Ordu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Study 1
Record Dates: First submitted 2019-02-06; First posted 2019-02-11 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Foot
Keywords: Foot Disease; Foot Care Protocol; Nursing Care
MeSH Terms: conditions — Foot Diseases

STUDY DESIGN:
Intervention Model Description: randomized-controlled trail
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- foot care protocol (Experimental): foot examination at the first interview, foot care and training once a month and weekly follow-up for 3 months, foot examination at the last interview (six month)
  Interventions: Other: foot care protocol
- Control (No Intervention): foot examination at the first interview, foot examination at the last interview (six month)

INTERVENTIONS:
Other: foot care protocol — foot assesment, foot care, foot care education
  Arms: foot care protocol

SUMMARY:
The study was carried out randomized-controlled experimental research to determine the foot health status and factors affecting it among elderly individuals, to develop a protective and developmental protocol for foot health of elderly individuals and to determine the effect of this protocol on foot health problems, foot care knowledge levels and foot care behaviors.

DETAILED DESCRIPTION:
Data for the foot health status and factors affecting it among elderly individuals were collected from 28 April 2017 to 5 February 2018. The population of the study comprised 132 elderly individuals living in Nursing Home linked to the Ministry of Family and Social Policies in Ordu Central County. In the research, 118 individuals in the nursing home were reached, the research began with 65 elderly individuals abiding by the inclusion criteria randomized into experimental and control groups and was completed with 57 individuals (experiment: 28, control: 29). Data were collected using the standardized mini mental test, elderly descriptive form, foot examination form, foot care knowledge level form, foot care behavior scale, falling form.. Ethics committee permission, organization permission and written informed consent from individuals were obtained. Five interviews were performed with elderly individuals in the experimental group, while only two interviews were held with elderly individuals in the control group to apply the data collection tools.

ELIGIBILITY:
Inclusion Criteria:

Living in nursing home during the research process, Not dependent on bed, Self-sufficient, No communication problem, Elderly people have good cognitive functions ,(According to the revised mini mental test) Elderly people with any foot problem (dermatological, orthopaedic, circulation, sensory problems, problems related to the feet, self-care problems),

Exclusion Criteria:

Elderly people who are diagnosed with Diabetes Mellitus

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 57 (Actual)
Dates: Start 2017-04-28 (Actual); Primary Completion 2017-06-16 (Actual); Study Completion 2018-02-05 (Actual)

PRIMARY OUTCOMES:
Change from foot examination questionnaire at baseline and sixth month | Baseline, 6th month
  This questionnaire was developed by the researchers and evaluated the foot health of elderly people. It contains 26 questions in three part section. This form enables the determination of the diseases / problems in the foot.
Change from foot care knowledge form at baseline and sixth month | Baseline, 6th month
  This form was developed by researchers and evaluated the level of knowledge of foot care. It contains 10 questions. This form evaluated on total score (minimum:0, maximum:10). Higher values represent a better outcome.
Change from foot self care observation guide at baseline and sixth month | Baseline, 6th month
  This scale evaluates the level of foot care behaviors of people. It contains 15 item. This scale evaluated on total score (minimum:15, maximum:75). Higher values represent a better outcome.
Change from falling questionnaire at baseline and sixth month | Baseline, 6th month
  This questionnaire was developed by the researchers and evaluated the number of elderly people.

CONTACTS AND LOCATIONS:
Overall Officials: Aslıhan Çatıker, Phd, Principal Investigator — Ordu University
Locations (1):
- Ahmet Cemal Mağden Nursing Home, Ordu, Altınordu, Turkey (Türkiye)